CLINICAL TRIAL: NCT05443958
Title: The Role of IEEG in the Localization of EZ and Its Relationship With Prognosis
Brief Title: The Role of Intracranial Electroencephalography (IEEG) in the Localization of Epileptogenic Zones (EZ) and Its Relationship With Prognosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-910
Record Dates: First submitted 2022-06-22; First posted 2022-07-05 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-06

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Seizure free group
- Not seizure free group

INTERVENTIONS:
Other:

SUMMARY:
The mechanism of epilepsy pathogenesis is complex and not fully defined, and about 20-30% of patients with seizures that cannot be completely controlled by drugs become drug-resistant epilepsy. For focal drug-resistant epilepsy, surgical removal of the epileptogenic zone can control seizures, but the overall seizure-free rate in the long term after surgery is 60-70%, and the results are still not satisfactory. Accurate assessment of the location and extent of the epileptogenic zone and its adequate excision are prerequisites for the success or failure of surgery. Intracranial EEG (iEEG) has been shown to be the most accurate method for determining the location and boundaries of the epileptogenic zone. It can selectively record the local cortical electrical activity through intracranial electrodes and achieve high temporal resolution for long-range recording, reliably reflecting the continuous dynamic changes of EEG during interictal and ictal periods. The in-depth analysis of iEEG can improve the efficacy of epilepsy surgery and provide important information to reveal the pathogenesis of epilepsy.

ELIGIBILITY:
Inclusion Criteria:

1. Complete clinical history;
2. IEEG monitoring at least one habitual seizure；
3. Follow up for at least 1 year；
4. Signed informed consent.

Exclusion Criteria:

1. Habitual seizures were not found in iEEG monitoring;
2. No operation was performed;
3. Lost to follow-up for various reasons within 1 year after surgery.

Ages: 3 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: We reviewed consecutive patients with drug-resistant focal epilepsy who underwent intracranial electroencephalography (IEEG) evaluation as well as resective surgery in our epilepsy centre. They were all followed-up for > 1 years after surgery. The patients had a comprehensive evaluation including detailed history, neuropsychological testing, neuroimaging study and video-EEG examination.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2023-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Comparison of clinical data and IEEG characteristics in the seizure-free and not seizure-free groups | 1-2 years
  Compare two groups of patients with clinical data (sex, age at onset, age at surgery, epilepsy duration, seizure lateralization/localization, MRI findings, Pathology) and EEG characteristics (contact number, EEG onset pattern, IEEG power of each frequency band, functional connectivity of each frequency band).

CONTACTS AND LOCATIONS:
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China, Hangzhou, China

IPD SHARING:
Plan to Share IPD: No